CLINICAL TRIAL: NCT00423462
Title: First Experimental Study of Transference Interpretations (FEST)
Brief Title: First Experimental Study of Transference-Interpretations (FEST)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: The Research Council of Norway (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FEST307/95
Record Dates: First submitted 2007-01-16; First posted 2007-01-18 (Estimated); Last update posted 2007-08-27 (Estimated); Status verified 2007-08

CONDITIONS: Mood Disorders; Anxiety Disorders; Personality Disorders
Keywords: Psychotherapy; Long-term effects
MeSH Terms: conditions — Mood Disorders; Anxiety Disorders; Personality Disorders

INTERVENTIONS:
Behavioral: Brief dynamic psychotherapy

SUMMARY:
Analysis of the ongoing patient-therapist interaction, the transference, is considered a key active ingredient in psychoanalytically oriented psychotherapy and psychoanalysis.However, one century after Sigmund Freuds's famous "Dora" case, the first clinical description of transference, no study of transference interpretations have been published.In the present study 100 out-patients were randomized to receive one year weekly dynamic psychotherapy, with and without transference interpretations. That is, one treatment component,transference interpretations, were added to a comparison condition, therapy of the same format, by the same therapists, but without use of transference interpretation.

All treatment session were audiotaped, and treatment integrity have been carefully checked. Patients were evaluated at treatment termination, one year after treatment termination and three years after treatment termination. Enrollment of patients started january 1993, and all follow-up evaluations completed by December 2005.

DETAILED DESCRIPTION:
This study is designed to measure specific long-term effects of transference interpretations in dynamic psychotherapy, using an experimental dismantling design. One hundred psychiatric out-patients, referred to seven study therapists, to receive exploratory dynamic psychotherapy, were randomized to one year weekly dynamic psychotherapy, with and without transference interpretations.They suffered from mood,anxiety,and personality disorders or interpersonal problems not due to a mental disorder. All treatment sessions were audiotaped and treatment integrity carefully checked.All patients have been evaluated before treatment, after treatment, one year after termination of treatment, and three years after termination of treatment. The main outcome measures were the Psychodynamic Functioning Scales (PFS) and Inventory of Interpersonal Problems-Circumplex version (IIP-C).Chang over time is assessed using linear mixed model analyses.

The main hypothesis is that patients treated with transference interpretations will have a more favourable course over the whole study period of four years.

The second hypothesis is that suitable patients, that is patients with a life long pattern of more mature object relations (QOR) and/or patients without comorbid personality disorders will do better with transference interpretations.

Insight and identification with the therapist will be analyzed as putative mediators of long-term change in interpersonal functioning

ELIGIBILITY:
Inclusion Criteria:

* Age 20 - 60 years
* Diagnoses Mood-disorder, non-psychotic
* Anxiety disorders
* Personality disorders
* Interpersonal problems not due to a mental disorder

Exclusion Criteria:

* Psychotic disorders
* Bipolar disorder
* Organic brain disorder
* Substance abuse
* Long-term (years) disability
* Mental retardation

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100
Dates: Start 1993-01; Study Completion 2005-12

PRIMARY OUTCOMES:
The Psychodynamic Functioning Scales (PFS), clinician rated
Inventory if Interpersonal Problems-Circumplex version (IIP-C), self-report

SECONDARY OUTCOMES:
The Global Assessment of Functioning Scale (GAF)
Global Severity Index (GSI) from SCL-90-R

CONTACTS AND LOCATIONS:
Overall Officials: Per Høglend, M.D. Ph. D., Principal Investigator — Department of Psychiatry, Faculty of Medicine, Unoversity of Oslo
Locations (1):
- Department of Psychiatry, Faculty of Medicine, University of Oslo, Oslo, Norway

REFERENCES:
- [Result] Hoglend P, Amlo S, Marble A, Bogwald KP, Sorbye O, Sjaastad MC, Heyerdahl O. Analysis of the patient-therapist relationship in dynamic psychotherapy: an experimental study of transference interpretations. Am J Psychiatry. 2006 Oct;163(10):1739-46. doi: 10.1176/ajp.2006.163.10.1739. PMID 17012684
- [Derived] Nissen-Lie HA, Dahl HJ, Hoglend PA. Patient factors predict therapists' emotional countertransference differently depending on whether therapists use transference work in psychodynamic therapy. Psychother Res. 2022 Jan;32(1):3-15. doi: 10.1080/10503307.2020.1762947. Epub 2020 May 13. PMID 32404003
- [Derived] Tallberg P, Ulberg R, Johnsen Dahl HS, Hoglend PA. Core conflictual relationship theme: the reliability of a simplified scoring procedure. BMC Psychiatry. 2020 Apr 6;20(1):150. doi: 10.1186/s12888-020-02558-4. PMID 32252696
- [Derived] Sorbye O, Dahl HJ, Eells TD, Amlo S, Hersoug AG, Haukvik UK, Hartberg CB, Hoglend PA, Ulberg R. Psychodynamic case formulations without technical language: a reliability study. BMC Psychol. 2019 Oct 24;7(1):67. doi: 10.1186/s40359-019-0337-5. PMID 31651367
- [Derived] Ulberg R, Ness E, Dahl HS, Hoglend PA, Critchfield K, Blayvas P, Amlo S. Relational interventions in psychotherapy: development of a therapy process rating scale. BMC Psychiatry. 2016 Sep 6;16(1):310. doi: 10.1186/s12888-016-1021-4. PMID 27600314
- [Derived] Ulberg R, Amlo S, Hoglend P. Manual for Transference Work Scale; a micro-analytical tool for therapy process analyses. BMC Psychiatry. 2014 Nov 18;14:291. doi: 10.1186/s12888-014-0291-y. PMID 25404145
- [Derived] Ulberg R, Amlo S, Hersoug AG, Dahl HS, Hoglend P. The effects of the therapist's disengaged feelings on the in-session process in psychodynamic psychotherapy. J Clin Psychol. 2014 May;70(5):440-51. doi: 10.1002/jclp.22088. Epub 2014 Mar 27. PMID 24677205
- [Derived] Ulberg R, Hoglend P, Marble A, Johansson P. Women respond more favorably to transference intervention than men: a randomized study of long-term effects. J Nerv Ment Dis. 2012 Mar;200(3):223-9. doi: 10.1097/NMD.0b013e318247cb6d. PMID 22373759
- [Derived] Hoglend P, Hersoug AG, Bogwald KP, Amlo S, Marble A, Sorbye O, Rossberg JI, Ulberg R, Gabbard GO, Crits-Christoph P. Effects of transference work in the context of therapeutic alliance and quality of object relations. J Consult Clin Psychol. 2011 Oct;79(5):697-706. doi: 10.1037/a0024863. PMID 21859184
- [Derived] Ulberg R, Hoglend P, Marble A, Sorbye O. From submission to autonomy: approaching independent decision making. A single-case study in a randomized, controlled study of long-term effects of dynamic psychotherapy. Am J Psychother. 2009;63(3):227-43. doi: 10.1176/appi.psychotherapy.2009.63.3.227. PMID 19845088
- [Derived] Ulberg R, Johansson P, Marble A, Hoglend P. Patient sex as moderator of effects of transference interpretation in a randomized controlled study of dynamic psychotherapy. Can J Psychiatry. 2009 Feb;54(2):78-86. doi: 10.1177/070674370905400205. PMID 19254438